CLINICAL TRIAL: NCT03885973
Title: Lactobacillus Plantarum IS 10560 Supplementation in Women With Functional Constipation: Molecular Profile of Fecal Microbiome With NGS Method
Brief Title: Lactobacillus Plantarum IS 10560 Supplementation in Women With Functional Constipation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fakultas Kedokteran Universitas Indonesia (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Murdani Abdullah, Clinical Professor, Fakultas Kedokteran Universitas Indonesia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18-01-0060
Record Dates: First submitted 2019-03-17; First posted 2019-03-22 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Constipation - Functional
Keywords: SCFA; Probiotic; Lactobacillus plantarum; Functional constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactobacillus plantarum (Experimental): 1 bottle of fermented milk (100 g) containing probiotic Lactobacillus plantarum IS-10506 1.0x10^8 CFU will be given daily for three weeks.
  Interventions: Drug: Lactobacillus plantarum
- Placebo (Placebo Comparator): 1 bottle of fermented milk (100 g) containing placebo will be given daily for three weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lactobacillus plantarum — Fermented milk containing probiotic Lactobacillus plantarum for three weeks
  Arms: Lactobacillus plantarum
Drug: Placebo — Fermented milk containing placebo for three weeks
  Arms: Placebo

SUMMARY:
In this study, the investigators measured the SCFA (Butyrate, Acetate and Propionate) as a Biomarker improvement symptom and quality of life women with functional constipation after supplementation of commensal bacterial fermented milk Lactobacillus plantarum (isolated from indigenous probiotics from Dadih, West Sumatra) for 21 days

ELIGIBILITY:
Inclusion Criteria:

* Being declared healthy based on initial examination and the Structured Interview Questionnaire (SIQ)
* Having the symptoms and signs of functional constipation refer to ROME IV
* Able to communicate well
* Able to consume 1 bottle of fermented milk each day for three weeks
* Not using antibiotic no later than one week before supplementation

Exclusion Criteria:

* Diagnosed with functional bowel disorder
* Using anesthesia at least 4 weeks before treatment
* Having a serious pathological disorder (carcinoma)
* During healing phase of acute gastrointestinal disorders at least 4 weeks before treatment
* Having severe heart disease
* Taking chronic medications such as antidepressants or analgesics

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2018-07-28 (Actual); Primary Completion 2018-08-22 (Actual); Study Completion 2018-08-22 (Actual)

PRIMARY OUTCOMES:
Short Chain Fatty Acid (SCFA) titer | Three weeks after intervention
  Short Chain Fatty Acid (SCFA) titer that will be analyzed by Gas chromatography-mass spectrometry (GCMS) consists of three metabolites:
  * Butyrate will be shown in mM unit measure, higher value represents better outcome
  * Acetate will be shown in mM unit measure, higher value represents better outcome
  * Proprionate will be shown in mM unit measure, higher value represents better outcome
Functional constipation symptom improvement (1) | Three weeks after intervention
  Functional constipation symptom improvement (1) will be measured by improvement of PAC Sym questionnaire score. PAC Sym (Patient Assessment of Constipation Symptoms) has a minimum score of 0, maximum score 48, lower value represents better outcome
Functional constipation symptom improvement (2) | Three weeks after intervention
  Functional constipation symptom improvement (2) will be measured by improvement of PAC QoL questionnaire score. PAC QoL (Patient Assessment of Constipation Quality of Life) has a minimum score of -20, maximum score 92, lower value represents better outcome
Molecular Profile of Fecal Microbiome | Three weeks after intervention
  Microbiome profile from faecal samples will be analyzed with NGS (Next Gen Sequencing) method. The result will be analyzed with MiSEq Reporter software (MSR) and will be presented in nM unit measure.

CONTACTS AND LOCATIONS:
Overall Officials: Pratiwi D Kusumo, Principal Investigator — Fakultas Kedokteran Universitas Indonesia
Locations (1):
- Puskesmas Petamburan, Jakarta, DKI Jakarta, Indonesia

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-29): https://cdn.clinicaltrials.gov/large-docs/73/NCT03885973/Prot_SAP_000.pdf